CLINICAL TRIAL: NCT05408065
Title: A Randomized Single-blinded Clinical Trial of the Efficacy of Intra-articular Infiltration of Cingal (Sodium Hyaluronate/Triamcinolone) Versus Cortisone (Triamcinolone) in Patients With Osteoarthritis of the Shoulder.
Brief Title: Comparison of the Analgesic Effect of 2 Shoulder Infiltrations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-10659
Record Dates: First submitted 2022-05-11; First posted 2022-06-07 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Infiltration; Shoulder Osteoarthritis
Keywords: infiltration; Osteoarthritis; hyaluronic acid
MeSH Terms: conditions — Osteoarthritis | interventions — triamcinolone hexacetonide; Hyaluronic Acid; Cortisone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cingal (Experimental): A single infiltration of Cingal, 4 mL, 88 of mg hyaluronic acid and 18 mg of triamcinolone hexacetonide
  Interventions: Drug: Triamcinolone Hexacetonide and hyaluronic acid
- Cortisone (Active Comparator): A single infiltration of cortisone, 40mg of triamcinolone and 4mL of bupivacaine 0.25%
  Interventions: Drug: Triamcinolone Hexacetonide

INTERVENTIONS:
Drug: Triamcinolone Hexacetonide and hyaluronic acid — infiltration under fluoroscopy
  Other Names: Cingal
  Arms: Cingal
Drug: Triamcinolone Hexacetonide — infiltration under fluoroscopy
  Other Names: Cortisone
  Arms: Cortisone

SUMMARY:
For patients suffering of osteoarthritis, only analgesic treatments such as anti-inflammatory drugs and cortisone infiltrations provide significant but temporary relief of their pain. The objective is to compare the analgesic effect of 2 infiltrations: Cingal (sodium hyaluronate and triamcinolone) versus cortisone (triamcinolone). It is anticipated that the Cingal infiltration will have a greater analgesic effect than a simple cortisone infiltration in patients with moderate to severe osteoarthritis of the shoulder.

Method:

* Randomized controlled trial
* Monocentric
* Randomization will be done using sealed envelopes

DETAILED DESCRIPTION:
Osteoarthritis is a degenerative joint disease. The progressive erosion of cartilage generates inflammation, pain, and progressive deterioration of joint mobility. Synthetic molecules similar to hyaluronic acid have made it possible to offer patients the option of visco-supplementation by intra-articular injection. It decreases inflammation and pain. CINGAL (Anika Therapeutics, Inc., Bedford, MA), which combines the lubricating action of hyaluronic acid and the anti-inflammatory action of triamcinolone hexacetonide, is one of the available treatments. Several studies have demonstrated the effectiveness of hyaluronic acid in the relief of gonarthrosis. However, the efficacy between an infiltration of hyaluronic acid combined with triamcinolone and a corticosteroid infiltration for glenohumeral osteoarthritis is hardly reviewed in scientific studies.

Primary objective: To compare the analgesic effect of two different infiltrations.

Secondary outcome: To evaluate the patient's functional ability

It is anticipated that a CINGAL infiltration will have a greater beneficial effect than a simple cortisone infiltration in patients with mild to severe shoulder OA.

84 patients with moderate to severe shoulder osteoarthritis will be recruited to receive intra-articular infiltration of CINGAL or cortisone. The infiltration will be randomly assigned. A standard x-ray and magnetic resonance imaging examination will be performed before the infiltration. Demographic data, medical history and 2 questionnaires will be completed prior to infiltration.

Once the evaluation is completed, the patient is randomized and referred to radiology to receive his infiltration under fluoroscopy by a radiologist assigned to the project. Two electronic questionnaires and a medication diary will be sent to the patient at 1, 3 and 6 months post-infiltration.

ELIGIBILITY:
Inclusion Criteria:

* A clinical examination that confirms the radiological diagnosis of moderate to severe primary shoulder osteoarthritis, stage II and above, according to the Samilson-Prieto classification.
* Patients aged between 20 and 90 years.
* A patient with bilateral shoulder osteoarthritis will choose the side of the infiltration, only one side can be chosen to participate in the study.
* The patient must have a clinical pain threshold of a minimum of 4/10 on the visual analogue scale.
* The patient must have the cognitive ability to read and fill out the questionnaires.
* The patient must be able to read and understand French or English

Exclusion Criteria:

* Presence of a transfixing rotator cuff tear assessed on MRI.
* No previous shoulder reconstruction surgery.
* Pregnant woman.
* A patient who has received a cortisone infiltration within 6 months prior to the start of the study.
* A patient who has received a platelet-rich plasma or a hyaluronic acid infiltration within 12 months prior to the start of the study.
* Diagnosis of avascular necrosis.
* Disease affecting the studied joint (systemic inflammatory disease, history of septic arthritis, osteonecrosis, etc.)
* Suspicion or presence of active local infectious process.
* Presence or suspicion of neoplasia or local metastasis.
* Severe trauma to the shoulder ( ≤ 3 months)
* Significant cognitive impairment or insufficient language proficiency to adequately answer the questionnaires.
* Any other serious medical condition that does not allow participation in the study or may be a contraindication to cortisone injection.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in VAS score | Change from baseline (preinfiltration visit) VAS score at 3 months after the infiltration
  Visual analogue score VAS; 0-10 scale, 0: no pain 10: worst possible pain

SECONDARY OUTCOMES:
Change in VAS score | Change from baseline (preinfiltration visit) VAS score at 1 month after the infiltration
  Visual analogue score VAS; 0-10 scale, 0: no pain 10: worst possible pain
Change in VAS score | Change from baseline (preinfiltration visit) VAS score at 6 months after the infiltration
  Visual analogue score VAS; 0-10 scale, 0: no pain 10: worst pain
Change in QuickDash disability/symptoms score | Change from baseline (preinfiltration visit) QuickDash score at 1 month after the infiltration
  QuickDash; 0-100 scale, 0: no difficulties 100: unable
Change in QuickDash disability/symptoms score | Change from baseline (preinfiltration visit) QuickDash score at 3 months after the infiltration
  QuickDash; 0-100 scale, 0: no difficulties 100: unable
Change QuickDash disability/symptoms score | Change from baseline (preinfiltration visit) QuickDash score at 6 months after the infiltration
  QuickDash; 0-100 scale, 0: no difficulties 100: unable
Change in QuickDash Work score | Change from baseline (preinfiltration visit) QuickDash score at 1 month after the infiltration
  QuickDash; 0-100 scale, 0: no difficulties 100: unable
Change in QuickDash Work score | Change from baseline (preinfiltration visit) QuickDash score at 3 months after the infiltration
  QuickDash; 0-100 scale, 0: no difficulties 100: unable
Change in QuickDash Work score | Change from baseline (preinfiltration visit) QuickDash score at 6 months after the infiltration
  QuickDash; 0-100 scale, 0: no difficulties 100: unable
Change in QuickDash Sport/Music score | Change from baseline (preinfiltration visit) QuickDash score at 1 month after the infiltration
  QuickDash; 0-100 scale, 0: no difficulties 100: unable
Change in QuickDash Sport/Music score | Change from baseline (preinfiltration visit) QuickDash score at 3 months after the infiltration
  QuickDash; 0-100 scale, 0: no difficulties 100: unable
Change in QuickDash Sport/Music score | Change from baseline (preinfiltration visit) QuickDash score at 6 months after the infiltration
  QuickDash; 0-100 scale, 0: no difficulties 100: unable

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Tétreault, MD FRCSC, Principal Investigator — CHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brox JI, Lereim P, Merckoll E, Finnanger AM. Radiographic classification of glenohumeral arthrosis. Acta Orthop Scand. 2003 Apr;74(2):186-9. doi: 10.1080/00016470310013932. PMID 12807327
- [Background] Hangody L, Szody R, Lukasik P, Zgadzaj W, Lenart E, Dokoupilova E, Bichovsk D, Berta A, Vasarhelyi G, Ficzere A, Hangody G, Stevens G, Szendroi M. Intraarticular Injection of a Cross-Linked Sodium Hyaluronate Combined with Triamcinolone Hexacetonide (Cingal) to Provide Symptomatic Relief of Osteoarthritis of the Knee: A Randomized, Double-Blind, Placebo-Controlled Multicenter Clinical Trial. Cartilage. 2018 Jul;9(3):276-283. doi: 10.1177/1947603517703732. Epub 2017 May 23. PMID 28535076
- [Background] Noel E, Hardy P, Hagena FW, Laprelle E, Goebel F, Faure C, Favard L, Gaudin P, Christ R, Baudot C, Dietl J, Goupille P. Efficacy and safety of Hylan G-F 20 in shoulder osteoarthritis with an intact rotator cuff. Open-label prospective multicenter study. Joint Bone Spine. 2009 Dec;76(6):670-3. doi: 10.1016/j.jbspin.2009.10.008. PMID 19945321
- [Background] He WW, Kuang MJ, Zhao J, Sun L, Lu B, Wang Y, Ma JX, Ma XL. Efficacy and safety of intraarticular hyaluronic acid and corticosteroid for knee osteoarthritis: A meta-analysis. Int J Surg. 2017 Mar;39:95-103. doi: 10.1016/j.ijsu.2017.01.087. Epub 2017 Jan 27. PMID 28137554
- [Background] Petrella RJ, Petrella M. A prospective, randomized, double-blind, placebo controlled study to evaluate the efficacy of intraarticular hyaluronic acid for osteoarthritis of the knee. J Rheumatol. 2006 May;33(5):951-6. PMID 16652426
- [Background] Petrella RJ, Emans PJ, Alleyne J, Dellaert F, Gill DP, Maroney M. Safety and performance of Hydros and Hydros-TA for knee osteoarthritis: a prospective, multicenter, randomized, double-blind feasibility trial. BMC Musculoskelet Disord. 2015 Mar 18;16:57. doi: 10.1186/s12891-015-0513-6. PMID 25887932
- [Background] Smith C, Patel R, Vannabouathong C, Sales B, Rabinovich A, McCormack R, Belzile EL, Bhandari M. Combined intra-articular injection of corticosteroid and hyaluronic acid reduces pain compared to hyaluronic acid alone in the treatment of knee osteoarthritis. Knee Surg Sports Traumatol Arthrosc. 2019 Jun;27(6):1974-1983. doi: 10.1007/s00167-018-5071-7. Epub 2018 Jul 25. PMID 30046992
- [Background] Samilson RL, Prieto V. Dislocation arthropathy of the shoulder. J Bone Joint Surg Am. 1983 Apr;65(4):456-60. PMID 6833319
- [Background] Tammachote N, Kanitnate S, Yakumpor T, Panichkul P. Intra-Articular, Single-Shot Hylan G-F 20 Hyaluronic Acid Injection Compared with Corticosteroid in Knee Osteoarthritis: A Double-Blind, Randomized Controlled Trial. J Bone Joint Surg Am. 2016 Jun 1;98(11):885-92. doi: 10.2106/JBJS.15.00544. PMID 27252432
- [Background] Walch G, Badet R, Boulahia A, Khoury A. Morphologic study of the glenoid in primary glenohumeral osteoarthritis. J Arthroplasty. 1999 Sep;14(6):756-60. doi: 10.1016/s0883-5403(99)90232-2. PMID 10512449
- [Background] Zhang B, Thayaparan A, Horner N, Bedi A, Alolabi B, Khan M. Outcomes of hyaluronic acid injections for glenohumeral osteoarthritis: a systematic review and meta-analysis. J Shoulder Elbow Surg. 2019 Mar;28(3):596-606. doi: 10.1016/j.jse.2018.09.011. Epub 2018 Nov 28. PMID 30502030